CLINICAL TRIAL: NCT03821961
Title: The Effect of Metabolic Surgery on the Endocrine Function of Pancreas: Clinical Value of 18F-FDOPA PET/CT Imaging
Brief Title: 18F-FDOPA PET/CT Imaging in Patients Undergoing Metabolic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Myungmoon Pharma. Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Sungsoo Park, Professor, Korea University Anam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STARDOM-PET
Record Dates: First submitted 2019-01-22; First posted 2019-01-30 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 2; PreDiabetes; Obesity
Keywords: Diabetes Mellitus, Type 2; PreDiabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metabolic surgery (Experimental): Roux-en-Y gastric bypass, Sleeve gastrectomy
  Interventions: Procedure: Metabolic Surgery

INTERVENTIONS:
Procedure: Metabolic Surgery — Roux-en-Y gastric bypass, Sleeve gastrectomy

SUMMARY:
The aim of the study is to compare the endocrine function of pancreas between pre and post metabolic surgery in patients with type 2 diabetes or prediabetes. The study will examine the endocrine function of pancreas using 18F-FDOPA PET/CT imaging and various biochemical laboratory tests

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes or prediabetes
* Body mass index >25.0 kg/m2
* Written informed consent

Exclusion Criteria:

* Diabetes induced by chronic pancreatitis or pancreas cancer
* Chronic glucocorticoid usage
* Significant coronary artery disease or cerebrovascular disease within the previous 3 months
* Uncompensated congestive heart failure
* Severe pulmonary disease defined as FEV1 < 50% of predicted value
* End stage renal disease on dialysis
* Acute infectious disease within the previous 3 months
* Pulmonary thromboembolism or thrombophlebitis within the previous 3 months
* History of cancer (except for basal cell skin cancer or cancer in situ)
* Prior gastrointestinal surgery (except for appendectomy or hemorrhoidectomy)
* Gastrointestinal disorders, malabsorptive disorders, or inflammatory bowel disease
* History of chronic liver disease (except for NAFLD/NASH)
* Psychiatric disorders including dementia, active psychosis, severe depression requiring > 2 medications, history of suicide attempts, alcohol or drug abuse within the previous 5 years

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Uptake value of 18F-FDOPA PET/CT from baseline | 6 months
  Standardized Uptake Value

SECONDARY OUTCOMES:
Change in Glycated Hemoglobin from baseline | 6 months
  percent change
Change in Fasting Plasma Glucose from baseline | 6 months
  percent change
Changes in c-peptide level from baseline | 6 months
  percent change
Changes in Insulinogenic index from baseline | 6 months
  (insulin30 min - insulinfasting)/(glucose30 min - glucosefasting)
Changes in HOMA-IR(homeostatic model assessment for insulin resistance) from baseline | 6 months
  (insulinfasting × glucosefasting)/405
Changes in Matsuda index from baseline | 6 months
  Insulin sensitivity indices obtained from oral glucose tolerance testing (Diabetes Care 22:1462-1470, 1999)
Change in Body Mass Index (BMI) from baseline | 6 months
  percent change
Change in Systolic Blood Pressure from baseline | 6 months
  percent change
Change in serum level of HDL cholesterol from baseline | 6 months
  percent change
Change in serum level of Triglycerides from baseline | 6 months
  percent change
Change in serum level of LDL cholesterol from baseline | 6 months
  percent change
Change in serum level of Total Cholesterol from baseline | 6 months
  percent change
Change in serum level of High-sensitivity C-reactive Protein | 6 months
  percent change
Change in number of diabetes medication from baseline | 6 months
  number of medication
Change in dosage of diabetes medication from baseline | 6 months
  Dosage of medication
Change in number of hypertension medication from baseline | 6 months
  number of medication
Change in dosage of hypertension medication from baseline | 6 months
  Dosage of medication
Change in number of dyslipidemia medication from baseline | 6 months
  number of medication
Change in dosage of dyslipidemia medication from baseline | 6 months
  Dosage of medication
Change in serum level of amino acid metabolites from baseline | 6 months
  glucose homeostasis and energy expenditure related metabolites
Change in BDI scores of questionnaire from baseline | 6 months
  Beck Depression Inventory(Score range, 0-68)(Higer values represent a worse outcome)
Change in HDRS scores of questionnaire from baseline | 6 months
  Hamilton Depression Rating Scale(Score range, 0-54)(Higer values represent a worse outcome)
Change in SF-36 scores of questionnaire from baseline | 6 months
  36 Item Short Form Survery(Scale for quality of life)(Higer values represent a worse outcome) (Score range for physical health, 0-400) (Score range for mental health, 0-400)
Change in IWQOL scores of questionnaire from baseline | 6 months
  Impact of Weight on Quality of Life(Score range, 31-155)(Higer values represent a worse outcome)
Change in MAQOL scores of questionnaire from baseline | 6 months
  Moorehead-Ardelt Quality of Life(Score range, -3 to 3)(Higer values represent a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Sungsoo Park, MD, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No